CLINICAL TRIAL: NCT05213299
Title: Investigate the Change in Facial Pain Threshold During Auricular Acupuncture in Healthy Volunteers: A Pilot Study
Brief Title: Investigate the Change in Facial Pain Threshold During Auricular Acupuncture in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bui Pham Minh Man (Other)
Responsible Party: Sponsor-Investigator, Bui Pham Minh Man, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FWA00023448
Record Dates: First submitted 2021-12-21; First posted 2022-01-28 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers
Keywords: Auricular Acupuncture
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: 2-arm crossover design, randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First auricular acupuncture, then sham acupuncture in left ear (Experimental): Participants are experienced two phases of our study. The first phase, participants are received auricular acupuncture at TF4, AT4, LO1, LO3 points in the left ear. The second phase, participants are received sham acupuncture at the same points. The facial pain threshold will be recorded before and after performing auricular acupuncture.
  Interventions: Procedure: AURICULAR ACUPUNCTURE; Other: PLACEBO
- First auricular acupuncture, then sham acupuncture in right ear (Experimental): Participants are experienced two phases of our study. The first phase, participants are received auricular acupuncture at TF4, AT4, LO1, LO3 points in the right ear. The second phase, participants are received sham acupuncture at the same points. The facial pain threshold will be recorded before and after performing auricular acupuncture.
  Interventions: Procedure: AURICULAR ACUPUNCTURE; Other: PLACEBO

INTERVENTIONS:
Procedure: AURICULAR ACUPUNCTURE — Auricular acupuncture is a method for diagnosing and treating physical and psychosomatic dysfunctions by stimulating a specific point in the ear. To conducting this intervention, the investigators use press tack needles to perform auricular acupuncture.
Other: PLACEBO — For this intervention, instead of needles, the investigators use four pieces of tape.

SUMMARY:
Background: The effects and biological mechanisms of auricular acupuncture on the human body have been increasingly observed in clinical and experimental studies, particularly the analgesic effects. Auricular acupuncture in the Shenmen, Nervous Subcortex, Jaw and Tooth groups has been shown in the Acupuncture 2 textbook of the Faculty of Traditional Medicine - University of Medicine and Pharmacy, Ho Chi Minh City and clinical studies to be effective in reducing facial pain.

This study aims to examine: (1) the change in facial pain threshold when performing auricular acupuncture in the acupoints of Shenmen (TF4), Nervous Subcortex (AT4), Jaw (LO3) and Tooth (LO1) on the left ear, (2) the change in facial pain threshold when performing auricular acupuncture in the acupoints of Shenmen, Nervous Subcortex, Jaw and Tooth on the right ear and (3) examining the unfavorable effects of the procedure.

DETAILED DESCRIPTION:
The effects and biological mechanisms of auricular acupuncture on the human body have been increasingly observed in clinical and experimental studies, particularly the analgesic effects. When the downward neurotransmitter pathway is activated, endogenous opioids (beta endorphins) are released, which inhibit pain perception. Furthermore, according to the gate control theory (spinal segmentation mechanism), auricular acupuncture aids in the activation of pain-suppressive stimuli by myelinated afferent fibers (Aβ), as opposed to stimuli with damage from poorly myelinated (Aδ) or unmyelinated (C) fibers. Besides, according to human physiology, the trigeminal nerve is involved in sensory control of the face, has a branching distribution to the skin of the pinna, and has afferent conduction of mechanical stimuli acting on it. Auricular acupuncture in the Shenmen, Nervous Subcortex, Jaw and Tooth groups has been shown in the Acupuncture 2 textbook of the Faculty of Traditional Medicine - University of Medicine and Pharmacy, Ho Chi Minh City and clinical studies to be effective in reducing facial pain.

This was the first study in Vietnam to investigate the effect of auricular acupuncture on the change in facial pain threshold during auricular acupuncture on acupoints such as Shenmen, Nervous Subcortex, Jaw and Tooth. The findings of the study can be used to supplement scientific evidence regarding the effects of auricular acupuncture in the treatment of clinical facial pain.

The investigators performed a randomized, controlled crossover experiments. A crossover study has two advantages over both a parallel study and a non-crossover longitudinal study. First, the influence of confounding covariates is reduced because each crossover patient serves as their own control. In a randomized non-crossover study it is often the case that different treatment-groups are found to be unbalanced on some covariates. In a controlled, randomized crossover designs, such imbalances are implausible (unless covariates were to change systematically during the study). Second, optimal crossover designs are statistically efficient, and so require fewer subjects than do non-crossover designs (even other repeated measures designs). In our study, the subjects are randomly assigned to two arms of the study which receive different treatments. A crossover trial has a repeated measures design in which each patient is assigned to a sequence of two treatments, one of which is auricular acupuncture, and a placebo test is performed on that volunteer a week later. Wilcoxon sign-rank test, paired T test and Pearson's chi-squared test were used for comparison of means.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 29 who are in good health.
* BMI ranging from 18.5 to 22.9 kg/m2 (classification of IDI & WPRO for Asians).
* Voluntarily consented to participate in the study, read, was thoroughly explained, and signed the consent form to participate in the study.
* Mental and physical well-being were assessed throughout the study period (on the Depression Anxiety and Stress Scale of 21 with a stress score of 15 points).
* Vital signs are within normal ranges:

Pulse: 60-100 pulses per minute Systolic blood pressure: 90 to 139 mmHg. Diastolic blood pressure: 60 to 89 mmHg. Temperature: 36.3-37.1 degrees Celsius. At rest, the breathing rate is 16 3 times per minute, and the SpO2 level is 92%.

- Volunteers have no other chronic medical conditions: Thyroid disease, autonomic neuropathy, hypertension, diabetes, respiratory diseases (asthma, pneumonia, chronic obstructive pulmonary disease, etc.) etc) by asking for medical history and medical history.

Exclusion Criteria:

* A feeling of fear or anxiety appeared immediately before the test (rated on the Depression Anxiety and Stress Scale of 21 with stress scores greater than or equal to 15 points).
* Use of stimulants such as alcohol, beer, coffee, and tobacco within 24 hours before the study.
* The auricular skin was examined with lesions (scars, lacerations, scratches, bites).

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the change of facial pain threshold when using auricular acupuncture and using sham acupuncture in the left ear in healthy volunteers by the multi-capacity digital force gage FDIX of Wagner Inc (Newton Unit of Measurement) | During procedure
  Evaluate the change of facial pain threshold when using auricular acupuncture and using sham acupuncture in the left ear in healthy volunteers by the multi-capacity digital force gage FDIX of Wagner Inc (Newton Unit of Measurement)

SECONDARY OUTCOMES:
Evaluate the change of facial pain threshold when using auricular acupuncture and using sham acupuncture in the right ear in healthy volunteers by the multi-capacity digital force gage FDIX of Wagner Inc (Newton Unit of Measurement) | During procedure
  Evaluate the change of facial pain threshold when using auricular acupuncture and using sham acupuncture in the right ear in healthy volunteers by the multi-capacity digital force gage FDIX of Wagner Inc (Newton Unit of Measurement)

OTHER OUTCOMES:
Examine the unfavorable effects during the procedure by using a questionnaire | During procedure
  Examine the unfavorable effects during the procedure by using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Ahn C. B., S. J. Lee, J. C. Lee, J. P. Fossion, A. Sant'Ana. A clinical pilot study comparing traditional acupuncture to combined acupuncture for treating headache, trigeminal neuralgia and retro-auricular pain in facial palsy. J Acupunct Meridian Stud. 2011;4(1): 29-43. 2011. De Salles-Neto F. T., J. S. de Paula, Jgaj Romero, C. M. Almeida-Leite. Acupuncture for pain, mandibular function and oral health-related quality of life in patients with masticatory myofascial pain: A randomised controlled trial. J Oral Rehabil. 2020;47(10): 1193-1201. Hou P. W., H. C. Hsu, Y. W. Lin, N. Y. Tang, C. Y. Cheng, C. L. Hsieh. The History, Mechanism, and Clinical Application of Auricular Therapy in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:495684. Iunes D. H., C. Chaves Éde, C. Moura Cde, B. Côrrea, L. C. Carvalho, A. M. Silva, et al. Role of Auriculotherapy in the Treatment of Temporomandibular Disorders with Anxiety in University Students. Evid Based Complement Alternat Med. 2015;2015:430143. Oliveri A. C., J. A. Clelland, J. Jackson, C. Knowles. Effects of auricular transcutaneous electrical nerve stimulation on experimental pain threshold. Phys Ther. 1986 Jan;66(1):12-6. Kaniusas E., S. Kampusch, M. Tittgemeyer, F. Panetsos, R. F. Gines, M. Papa, et al. Current Directions in the Auricular Vagus Nerve Stimulation I - A Physiological Perspective. Front Neurosci. 2019 Aug 9;13:854.